CLINICAL TRIAL: NCT01605565
Title: Analyse Fonctionnelle Par Imagerie Dynamique de l'épithélium Respiratoire Chez Des Nourrissons Atteints de Mucoviscidose
Brief Title: Functional Analysis by Dynamic Imaging of the Respiratory Epithelium in Infants With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C11-01; 2011-A00384-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-04-11; First posted 2012-05-25 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: A nasal brushing — A nasal brushing in every nostril

SUMMARY:
Cystic fibrosis (CF) is characterized by airway inflammation and infection leading to progressive destruction of lungs. One of the most important abnormalities in CF is an abnormal processing of the mutated CFTR protein through the endoplasmic reticulum that causes abnormal location or even absence of the protein at the apical plasma membrane of airway epithelial cells. This abnormality results in a marked dehydration of the airway surface fluid, decreased mucus transport and airway obstruction. Nevertheless, the events that occur very early during the progression of the disease at the airway level in infants are not known. At cellular level, it has also been reported that the CFTR expression and localization could be related to the differentiation state of the airway epithelium. Furthermore, it has been reported that gap junctions could be involved in dysregulate inflammation process. In CF infants, many answers are still lacking. For a better understanding of the early stages of cystic fibrosis, it is of major interest to study respiratory epithelial cells obtained as early as possible. In 15 CF infants and 15 control infants, a nasal brushing will be performed by means of a soft sterile cytology brush. Samples will be used for cytological and functional studies: ciliary beating frequency, cAMP-dependent chloride efflux, potassium efflux, tight and gap junctions functionalities. These studies will be done in basal conditions and will be repeated after activation of the nasal epithelial cells by the bacteria, such as Staphylococcus aureus, which can be found very early in the course of CF disease.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is characterized by airway inflammation and infection leading to progressive destruction of lungs. One of the most important abnormalities in CF is an abnormal processing of the mutated CFTR protein through the endoplasmic reticulum that causes abnormal location or even absence of the protein at the apical plasma membrane of airway epithelial cells. This abnormality results in a marked dehydration of the airway surface fluid, decreased mucus transport and airway obstruction. Nevertheless, the events that occur very early during the progression of the disease at the airway level in infants are not known. At cellular level, it has also been reported that the CFTR expression and localization could be related to the differentiation state of the airway epithelium. Furthermore, it has been reported that gap junctions could be involved in dysregulate inflammation process. In CF infants, many answers are still lacking.

Is inflammation present before infection? Is native epithelium of CF infants more sensitive than controls? Could the investigators analyse the localisation and functionality of CFTR, tight and gap junctions in respiratory epithelial cells in CF infants? Could the activation of the epithelial cells by bacteria alter their functional properties? For a better understanding of the early stages of cystic fibrosis, it is of major interest to study respiratory epithelial cells obtained as early as possible. Although bronchoalveolar lavage has been proposed for this purpose, nasal brushing, which is a much less invasive technique, has seldom been used in CF infants. the investigators have shown that, by means of a simple nasal brushing technique easily performed and well tolerated, it is feasible, in infants, to harvest native respiratory cell sheets in order to analyse the airway epithelium functionality. In 15 CF infants and 15 control infants, a nasal brushing will be performed by means of a soft sterile cytology brush. Samples will be used for cytological and functional studies: ciliary beating frequency, cAMP-dependent chloride efflux, potassium efflux, tight and gap junctions functionalities. These studies will be done in basal conditions and will be repeated after activation of the nasal epithelial cells by the bacteria, such as Staphylococcus aureus, which can be found very early in the course of CF disease.

the investigators believe that the present study could help to understand the pathophysiology on the very early stages of CF disease.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis

Exclusion Criteria:

* > 6 months old
* Other respiratory disease
* Other allergic disease
* Other infectious disease: fever (> 38° C), respiratory distress
* Altered general health state, rash,

Ages: 1 Week to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2013-09-18 (Actual); Study Completion 2013-09-18 (Actual)

PRIMARY OUTCOMES:
The main objective is to analyze the functionality of the respiratory epithelium in CF infant using a nasal brushing technique: ciliary beating frequency, cAMP-dependent chloride efflux, potassium efflux, tight and gap junctions functionalities. | no time frame
  In 15 CF infants and 15 control infants, a nasal brushing will be performed by means of a soft sterile cytology brush. Samples will be used for cytological and functional studies: ciliary beating frequency, cAMP-dependent chloride efflux, potassium efflux, tight and gap junctions functionalities.

CONTACTS AND LOCATIONS:
Overall Officials: Michel ABELY, Professor, Principal Investigator — CHU REIMS
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Background] Mosler K, Coraux C, Fragaki K, Zahm JM, Bajolet O, Bessaci-Kabouya K, Puchelle E, Abely M, Mauran P. Feasibility of nasal epithelial brushing for the study of airway epithelial functions in CF infants. J Cyst Fibros. 2008 Jan;7(1):44-53. doi: 10.1016/j.jcf.2007.04.005. Epub 2007 Jun 5. PMID 17553758